CLINICAL TRIAL: NCT06614036
Title: Remimazolam Versus Midazolam for Sedation During Upper GI Endoscopy: a Randomized Controlled Trial
Acronym: REST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Koen Munters (Other)
Collaborators: Gelre Hospitals (Other); Rijnstate Hospital (Other)
Responsible Party: Sponsor-Investigator, Koen Munters, Prof. dr. B.L.A.M. Weusten, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REST-study; 2024-516432-94-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Sedation for Diagnostic Gastroscopy
Keywords: sedation; remimazolam; midazolam; gastroscopy; procedural sedation
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): Byfavo 20 mg powder for solution for injection, remimazolam. Each vial contains remimazolam besylate equivalent to 20 mg remimazolam. Concentration after reconstitution: 2.5 mg/ml.
  Interventions: Drug: Remimazolam
- Midazolam (Active Comparator): Midazolam 1mg/ml, solution for injection / infusion. Each 5ml ampoule contains 5mg midazolam. Concentration: 1mg/ml.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam — Byfavo 20 mg powder for solution for injection, remimazolam. Each vial contains remimazolam besylate equivalent to 20 mg remimazolam. Concentration after reconstitution: 2.5 mg/ml.
  Other Names: Midazolam
  Arms: Remimazolam
Drug: Midazolam — Midazolam 1mg/ml, solution for injection / infusion. Each 5ml ampoule contains 5mg midazolam. Concentration: 1mg/ml.
  Other Names: Remimazolam
  Arms: Midazolam

SUMMARY:
Rationale Midazolam is known for its safety, effectiveness for procedural sedation during gastrointestinal (GI) endoscopy and is used as standard sedative by endoscopists worldwide. Remimazolam is a novel, recently approved sedative, with the potential to facilitate a faster (neuropsychiatric) recovery. Therefore, it may potentially enable earlier discharge and improvement of post-procedural memory compared to midazolam. Furthermore, remimazolam may enhance patient satisfaction.

Objective The investigators aim to compare the use of remimazolam and midazolam for sedation during diagnostic upper GI endoscopies in a randomized clinical trial.

Main trial endpoints Time to full alertness (time interval from the last dosage midazolam or remimazolam to the first of 3 consecutive MOAA/S scores of 5).

Secondary trial endpoints Interval between arrival in the recovery room and full alertness, patient satisfaction (based on questionnaire after discharge and after 1 day), duration of amnesia (based on memory test after 1 day), time interval between last dosage of sedative and readiness for discharge (first Aldrete score of at least 9), total dosage and number of boluses for adequate sedation, time interval between first dosage of sedative and start of the procedure, endoscopist satisfaction (scored 0-10 after the procedure).

Trial design Randomized, multicenter, double blind, clinical trial, which will take 2 days for study participants.

Trial population Adult patients scheduled for diagnostic upper GI endoscopy with sedation. The anticipated use of fentanyl or other opioids during endoscopy is an exclusion criterium (n=148 patients).

Interventions Participants will be randomly assigned to receive either remimazolam or midazolam as a sedative and will be followed up until one day after the procedure. One group will receive midazolam as a sedative, and another group will receive remimazolam as a sedative. Both agents will be administered in accordance with current guidelines. Vital signs, MOAA/S scores, and Aldrete scores will be monitored. Additionally, a memory test and a questionnaire will be administered to the participants.

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks This study aims to evaluate two procedures employed in regular daily care. Both sedatives used in this study are considered safe and effective for procedural sedation. Therefore, the investigators anticipate minimal risk for the participants involved in the study. Participants will not be subjected to any additional interventions or hospital visits apart from randomization, data collection, and two short questionnaires to evaluate amnesia and patient satisfaction. There will be no direct benefits for the participants as a result of their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years.
* Scheduled for a diagnostic upper GI endoscopy with procedural sedation.
* Ability to provide written informed consent, and to understand the responsibilities of trial participation.

Exclusion Criteria:

* Anticipated use of opioids, such as a therapeutic endoscopy or any other reason.
* ASA score of 4.
* Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to full alertness | From last dosage of the sedative until full alertness, assessed up to 60 minutes after last dosage
  Time to full alertness, defined as the time interval from the last dosage of the sedative and full alertness. Full alertness is evaluated using the well-known and validated MOAA/S score. This score is developed and validated to measure the level of alertness in subjects who are sedated. Full alertness is defined as the first of 3 consecutive MOAA/S scores of at least 5.

SECONDARY OUTCOMES:
Patient satisfaction | From first administration sedative until 1 day after diagnostic endoscopy
  Patients satisfaction is scored using two different parts of a questionnaire modified from the patient satisfaction with sedation instrument (PSSI). The PSSI is a validated score of procedural sedation satisfaction for outpatient endoscopies. The complete PSSI includes 19 multiple choice type questions which are categorised into 4 sub-scales for describing a patient's satisfaction. In this study the investigators focused on the PSSI sub-scores for global satisfaction and procedural recall in a modified PSSI.
Post-sedation amnesia | From full alrtness until 1 day after diagnostic endoscopy
  Post-sedation amnesia is scored using a self-developed amnesia test.
Incidence adverse events | From first dosage of sedative until one day after diagnostic gastroscopy
  Incidence of adverse events related to midazolam and remimazolam.
Time interval between patient arrival in the recovery room and full alertness. | From arrival recovery room until full alertness, assessed up to 90 minutes after arrival in the recovery room
  Time interval between patient arrival in the recovery room and full alertness.
Endoscopist satisfaction | From first dosage of sedative until end of endoscopic procedure, assessed up to 15 minutes after end of endoscopic procedure
  Endoscopist satisfaction is scored by the endoscopist directly after the procedure (range 0-10, with 0 being the lowest score, and 10 the highest).
Time to readiness for discharge | From last dosage of sedative until readiness for discharge, assessed up to 90 minutes after last dosage
  Time to readiness for discharge, defined as the time interval from the last dosage of the sedative to readiness for discharge. Readiness for discharge is evaluated using the well-known and validated Aldrete score. This score is developed to measure when the patient recovery is sufficient for the patient to be discharged home. Readiness for discharge is defined as the first Aldrete score of at least 9.
Succes rate of sedation | From first dosage of sedative until end of endoscopic procedure, assesed up to 15 minutes after end of endoscopic procedure
  The success rate of sedation, defined as the percentage of procedures which will be finished as intended without requirement of > 5 boluses of midazolam and remimazolam, and without requirement for an alternative sedative.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Gelre Hospitals, Apeldoorn, Gelderland
  - Rijnstate hospital, Arnhem, Gelderland
  - St Antonius hospital, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are currently discussing this topic